CLINICAL TRIAL: NCT05154500
Title: Evaluating Iron and Zinc Bioavailability From Biofortified Potatoes to Reduce Malnutrition in the Andean Highlands
Brief Title: Iron and Zinc Bioavailability From Biofortified Potatoes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigacion Nutricional, Peru (Other)
Collaborators: Quadram Institute Bioscience (Other); University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: BB/S014039/1
Record Dates: First submitted 2021-11-19; First posted 2021-12-13 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Biofortification; Potato
Keywords: Biofortification; Zinc; Iron; Potato

STUDY DESIGN:
Intervention Model Description: Double blind randomized trial of naturally biofortified with iron or zinc potatoes to be carried out in Huancavelica.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofortified Potato with iron or zinc ('A') (Experimental): Women volunteers will consume biofortified ('A') for one day in zinc study, and 10 days in iron study Zinc study and a local non-fortified Peruanita potato variety ('B') in a randomized order (either A-B or B-A). The potatoes have significantly different (p<0.001) content of iron or zinc, but no significant differences in vitamin C or phenolics (p>0.05). Based on this study design, every woman is her own control.
  Interventions: Other: Iron biofortified potato; Other: Zinc biofortified potato
- Non Biofortified potato with iron or zinc ('B') (Placebo Comparator): Women volunteers will consume no biofortified ('B') for one day in zinc study, and 10 days in iron study
  Interventions: Other: Iron biofortified potato; Other: Zinc biofortified potato

INTERVENTIONS:
Other: Iron biofortified potato — A non-blinded randomized cross-over design with multiple meal feedings will be used to quantify iron bioavailability from iron biofortified and non-biofortified potatoes. Women volunteers will consume biofortified ('A') and a local non-fortified Peruanita potato variety ('B') in a randomized order (either A-B or B-A). The potatoes have significantly different (p<0.001) content of iron or zinc, but no significant differences in vitamin C or phenolics (p>0.05). Based on this study design, every woman is her own control.
Other: Zinc biofortified potato — A crossover study will be used to compare zinc bioavailability of biofortified and non-fortified potatoes. Nutritional pre-screening is not required as there are no major systemic influences on zinc absorption.Volunteers will be randomly assigned to consume first either the biofortified or the non-biofortified potato, and consume the second potato-type 30 days later. Zinc absorption from two meals of biofortified or non-fortified potato will be measured using the double stable isotope technique.

SUMMARY:
Two of the most common nutritional deficiencies are anemia and zinc deficiency. One strategy for combating nutritional deficiencies is biofortification. The primary objective of the proposed research is to determine in humans the bioavailability of iron and zinc from biofortified potatoes as compared to a non-fortified local variety. The secondary objective is to use the data obtained from the human studies to model the potential impact of the introduction of biofortified potatoes to the alleviation of iron and zinc deficiencies in the Andean Highlands and low and middle-income countries elsewhere.

Iron bioavailability studies: The investigators will compare bioavailability of iron from a non-fortified potato variety with a biofortified potato that has significantly higher iron content though the use of a randomized cross-over intervention study. Female volunteers will consume both biofortified potato extrinsically labelled with 58FeSO4 and a nonfortified potato labelled with 57FeSO4. Thirty women with marginal iron status (plasma ferritin < 25 ng/ml) will be selected from an initial screening of 180 women. Every woman will receive 2 different types of test meals in a series of 20 servings for 10 days each. Blood samples will be collected during screening and on days 1, 15, 26 and 40 and the amount of 58Fe and 57Fe incorporated into hemoglobin and serum ferritin quantified.

Zinc bioavailability study: The investigators will compare bioavailability of zinc from a non-fortified potato variety with that of a biofortified potato that has significantly higher zinc content (p<0.001) with a crossover study. Forty volunteers will be randomly assigned to receive first either the biofortified or the non-fortified potato and receive the second meal 30 days later. Zinc absorption from two meals will be measured using the double stable isotope technique. Every volunteer will be given an i.v. infusion of 70zinc and two test meals of 250 g cooked potato labelled extrinsically with 67zinc separated by 3-4 hr. A spot urine sample will be collected 96 hours after each set of test meal and the ratio of the two isotopes measured to calculate absorption of zinc from the test meal.

Modelling and Impact assessment: Data on bioavailability will be used in a Disability Adjusted Life Year model to assess the potential impact of biofortified potatoes to alleviate iron and zinc deficiencies in the Andean Highlands and low and middle-income countries elsewhere.

DETAILED DESCRIPTION:
Type of Study and population Double blind randomized trial of naturally biofortified potatoes to be carried out in Huancavelica, Perú. It will be recruited about 100 women and 80 men aged 18-45 years living in the city of Huancavelica.

ETHICS Applications was submitted and approved by Research Ethics Committee (REC) of the University of East Anglia Faculty of Medicine and Health (FMH) in Norwich (UK) and a REC of the Instituto de Investigacion Nutricional (IIN) in Peru.

Every participant will be fully informed of all the procedures and will be given the opportunity to ask questions and receive any further details participants require.

The procedures (blood samples, urine samples, anthropometry, dietary recall) will be explained to the individuals who agree to take part in the initial screening, and participants will be invited to sign the first consent form.

SPECIFIC METHODS FOR IRON STUDY (Phase 1) Sample size The study requires an enrollment of a total of 30 women to allow for 33% who do not adhere to the protocol, to reach a final sample size of 20 women. The investigators estimate that the investigators may need to screen about 100 women.

Nutritional Status As part of the screening all the potential candidates will be weighed and measured using standardized equipment.

Measurement of physical activity All the participants will be asked to use an actigraph (a tri-axial accelerometer) which measures physical activity (movement) in three dimensions.

Blood sample An appropriately trained member of the study team will collect a venous blood sample (approximately 6ml in a test tube with heparin) to measure ferritin, hemoglobin, and CRP (screening and 3 more times: baseline, 16 and 40 days after first day of potato intake).

Urine sample Participants will be asked to provide a urine sample (30ml) to carry out a pregnancy test using a test strip.

Sociodemographic and Food security survey The investigators will include a socioeconomic survey and the ELCSA food security questionnaire both will be applied to all enrolled participants.

Study Procedures According to the results of the screening and revision of the criteria for inclusion and exclusion and following information and verification that participants understand the iron study consent form, subjects will be invited to participate. Consented participants will be randomly assigned to consume one or other of the two types of potato (biofortified-A or not-B). The first potato variety will be given during the first 2 weeks (day 1-12) and the second sequence between days 15-26, (in both cases excluding weekend days Saturday and Sunday). The potatoes will be cooked in water and offered mashed.

Blood samples will be taken on 5 occasions, 1) at screening to verify compliance with the exclusion and inclusion criteria; then on day 1 before participants eat the first type of potato, day 15 before eating the second type of potato, day 26 after eating all both potato types and on day 40 two weeks after eating all the potato.

Consumption of the potato Each participant will be served 500 g of potato divided into two portions of 250 g each. each participant will take, depending on their allocation, 0.3 mg of 57FeSO4 (Peruanita potato) or 0.3 mg of 58FeSO4 (biofortified potato), diluted in 50 ml of distilled water, which should be drunk while participants are eating the potato - halfway through the meal. In addition, each participant will receive 200 ml of distilled water to drink. The isotopes will be provided by ETH (Swiss Federal Institute of Technology in Zurich). In addition, the isotopes that the investigators will use are stable isotopes, that is participants exist naturally in the environment and as such do not pose any risk.

Collection of biological samples for the measurement of iron using stable isotopes Blood samples will be collected throughout the intervention period as previously described and will be sent to ETH, Zurich, following standard operating procedures. Participants will be informed and will provide consent for the transfer and use of their samples outside Peru' for the purpose of this research study. Samples will be anonymized and will not be transported with personal identifiable data.

In terms of processing, samples will be mixed with NO3 and H2O2 and digested in a microwave, followed by separation of the iron from the blood matrix by way of exchange-anion chromatography and a solvent (diluent) or extraction from the solvent using distilled.

The isotopes will be analyzed using a plasma coupled inductive multicollector mass spectrometer (Neptune; Thermo Finnigan). The amount of the labelled iron isotopes 57Fe and 58Fe will be measured 14 days after consumption of both types of potato has been completed. The calculation (of absorption) will be done considering the subjects estimated blood volume based on weight, height, and the subject's measured hemoglobin concentration (considering the average of the initial and final blood sample). The calculation is based on the principle of isotopic dilution considering as the factor for the iron isotope marker rather than the monoisotopic marker8. For the calculation of the fraction absorbed the investigators will assume 80% incorporation of the absorbed iron.

SPECIFIC METHODS FOR ZINC STUDY (Phase 2) Sample size The study requires a samples size of 40 women. This allows for a 40% loss to reach a final total of 24 women.

Procedures According to the results of screening, and after checking that participants comply with all the inclusion criteria and none of the exclusion criteria participants will be invited to participate in the zinc part of the study. For this participant will be given the second consent form to read and those who accept and sign the form will be invited to participate in the study.

The people who accept will be randomly allocated to eat one or other of the types of potato (biofortified-A or no-B). All the participants will be given both types of potato but in different order, in this way each participant will be their own control. The first variety of potato will be given on day 1, after acceptance of participating in the study, and after accepting and signing the consent form for this part: (consumption protocol and second variety will be eaten 29 days after (the order of potato varieties will be randomly assigned).

The investigators will take blood samples on three occasions: enrolment and days 1 and 29 (the days when participants eat the potato) after fasting for 8 hours (food) and 6 hours (liquids).

Study Measurements Anthropometry As part of the screening all the potential candidates will be weighed and measured using standardized equipment. According to their weight and BMI the investigators will decide whether participants are eligible.

Consented participants will be asked to provide a venous blood sample (approximately 10ml in a test tube with heparin). Plasma and packed red cells will be obtained from the blood samples and stored at <18oC.

Urine sample Consented participants will provide a urine sample (30ml) as part of the screening phase to carry out a pregnancy test. On days 1, 3, 4, 5, 6, 7, 29, 32, 33, 34, 35 and 36 the investigators will collect urine samples to analyze zinc content. On each day the investigators need 100ml of urine, collected in the morning (between 7-12 o'clock in the morning).

Consumption of the potato The subjects will be given a total of 1000 g of potato in two 500 g portions. The first portion will be given while participants are fasted, (at least 8 hours for food and 6 hours for drink) and in two separate servings (each one 250 g). When participants have eaten the first 250 g serving, the subject will receive 0.25 mg of 67Zn diluted in 50 ml of bottled water and then participants will receive the second serving of potato. Two hours later, participants will receive an intravenous infusion of 70Zn (200 ug) diluted in 50 ml of bottled water. After a further 2 hours participants will receive the second two servings of potato, and, as before, after the first serving participants will receive 0.25 mg of 67Zn diluted in 50 ml of bottled water. During this period and for 3 hours after the second portion of potato the subject will not consume any food or liquid, except for water which participants will be provided with. Each subject will receive 200 ml of water with each meal and 200 ml of water between meals. Currently, using isotopes is the best method for measuring the absorption of zinc. In addition, the isotopes that will be used are stable isotopes, that is participants exist naturally in the environment and pose no risk. No food or drink can be consumed for at least 3 hours after eating the final portion of potato.

Blood samples for measurement of zinc The investigators will take a total of three blood samples in total. Absorption using stable isotopes (Day 29) The blood samples that have been collected will be sent to ETH, Zurich. ETH will undertake the analysis of CRP for Zinc. The CRP will be measured using an ELISA kit. The plasma zinc concentration will be measured by induction plasma coupled mass spectrometry.

Urine samples for measurement of zinc using stable isotopes Samples of urine will be concentrated using freeze drying and then mineralized by digestion in a microwave oven (MLS-Turbowave; MLS GmbH) using a mixture of HNO3 and zinc isolated from the master matrix by ion exchange chromatography. The investigators will use ultrapure acids for the preparation of the samples.

Determination of zinc absorption Blood and zinc isotopic composition will be analyzed in duplicate at the ETH Human Nutrition Laboratory. Urine samples will be mineralized by microwave digestion (MLS-ETHOS plus; MLS GmbH) using a mixture of HNO3 and H2O2 and zinc isolated from the sample matrix by ion-exchange chromatography (Wegmuller et al 2014). All acids used for the preparation of samples will be ultrapure. 70Zn:66Zn and 67Zn:66Zn isotopic ratios will be measured to determine 70Zn and 67Zn enrichment in the urine samples by using a high-resolution double-focusing magnetic sector field multi-collector inductively coupled plasma mass spectrometer (Finnigan Neptune; Thermo Electron).12 Fractional absorption of the 67Zn dose from the test meals will be calculated by using the oral to i.v. tracers ratio method applied to spot urine samples, according to principles described by Friel et al.

7-day food record Using the method of registering all foods eaten over a 7-day period the investigators can obtain information on all foods eaten in a week (including Saturday and Sunday). To achieve this, the investigators will ask the subjects to make a record of all foods consumed, details of food preparation, and all drinks (including water) that participants have eaten or drunk. Participants should note the meal at which the food and drink were consumed, and the time taken to eat it (breakfast, lunch, supper and between meals (snacks) and the amount eaten at each time of the day. To do this the investigators will give the subjects a tablet in which to register the consumption/meals and as well take a photo of all the food eaten.

METHODS SPECIFIC FOR IMPACT ASSESSMENT The data on dietary intake, serum ferritin and iron bioavailability will be used for two modelling approaches. Firstly, the investigators will apply the Disability Adjusted Life Year (DALY) method, which is an appropriate method to estimate nutritional and health impacts of biofortified crops. This will build upon models that have been developed jointly by CIP and IIN that has made assumptions concerning iron and zinc bioavailability from potatoes. Secondly, the investigators will use data on habitual iron intake, serum ferritin concentrations and calculated physiological requirements for iron to adapt a model estimate dietary iron bioavailability in Europe, the Andean highland region and, more generally, to low- and middle-income countries.

ELIGIBILITY:
INCLUSION CRITERIA FOR IRON PART:

Inclusión Criteria:

* Healthy women aged 18-45 years
* Marginal levels of iron in blood as measured by serum ferritin <25ug/L.
* BMI: 18.5 to 25 kg/m2.
* Body weight <65kg.
* Prepared to attend study visits at the investigator site over a period of approximately 4 weeks (total 20 days) and, eat each day the prepared potatoes and then stay for a further 3 hours after eating the potato.
* Able to understand study requirements and provide written informed consent.

Exclusion criteria

* Severe anaemia (Hb<80g/L)
* Evidence of inflammation as measured by C-reactive protein (CRP) (>5mg/100ml).
* Gastrointestinal or renal problems; self-reported metabolic disease based on prior diagnosis, or a prior screening questionnaire.
* Pregnancy (positive urine test).
* Currently breastfeeding.
* Currently taking any medication, antibiotic or supplement that might be expected to affect iron metabolism.
* Not willing to discontinue taking iron supplements for at least 2 weeks before taking part in the study.
* No significant blood loss in the last 6 months due to trauma, major surgery or blood donation.
* Not able to eat the full amount of the potato.
* Allergy to any ingredients of the test meal.

INCLUSION CRITERIA FOR ZINC PART:

Inclusion Criteria:

* Healthy women aged 18-45 years.
* BMI 18.5-25 kg/m2.
* Willing to come to the study centre to eat the prepared potatoes on two occasions with a wash-out of 30 days (each day a different variety of potato) and to remain in the study centre for 7-8 hours in both occasions (one day to eat the biofortified variety and the other day the common variety) and as well to comply with all the study processes.
* Able to understand the consent form and to sign it.

Exclusion criteria

* Severe anaemia (Hb<80g/dL adjusted for altitude).
* Inflammation measured as CRP (>5mg/100ml).
* Gastrointestinal, renal problems, metabolic illness (self-reported or prior diagnosis or evident from replies in a questionnaire).
* Pregnant (urine test).
* Breastfeeding.
* Taking medication, antibiotic or supplement that could affect zinc metabolism.
* Not willing to discontinue supplements for at least 2 weeks before participating in the study.
* Significant blood loss in the last 6 months due to trauma, surgery or blood donation.
* Unable to eat all the potato.
* Allergy to any ingredients of the test meal.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 179 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2021-11-30 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Percent of iron absorption from a biofortified potato vs non-biofortified potato | 40 days
  Percent of of iron absorption from a biofortified potato is higher as compared to a non-fortified local variety.

SECONDARY OUTCOMES:
Percent of zinc absorption from a biofortified potato vs non-biofortified potato | 35 days
  Percent of of zinc absorption from a biofortified potato is higher as compared to a non-fortified local variety.

CONTACTS AND LOCATIONS:
Overall Officials: Reyna Liria-Domínguez, PhD, Principal Investigator — Instituto de Investigación Nutricional
Locations (2):
- Peru (2):
  - International Potato Center, Lima
  - Research Nutritional Institute, Lima

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liria-Dominguez R, Penny M, Kroon PA, Burgos G, Dainty J, Zeder C, Zimmermann MB, King J, Mithen R, Boy E, Al-Jaiballi O, Fairweather-Tait S. Biofortified Yellow-Fleshed Potatoes Provide More Absorbable Zinc than a Commonly Consumed Variety: A Randomized Trial Using Stable Isotopes in Women in the Peruvian Highlands. J Nutr. 2023 Oct;153(10):2893-2900. doi: 10.1016/j.tjnut.2023.08.028. Epub 2023 Aug 28. PMID 37648112
- [Derived] Burgos G, Liria R, Zeder C, Kroon PA, Hareau G, Penny M, Dainty J, Al-Jaibaji O, Boy E, Mithen R, Hurrell RF, Salas E, Zum Felde T, Zimmermann MB, Fairweather-Tait S. Total Iron Absorbed from Iron-Biofortified Potatoes Is Higher than that from Nonbiofortified Potatoes: A Randomized Trial Using Stable Iron Isotopes in Women from the Peruvian Highlands. J Nutr. 2023 Jun;153(6):1710-1717. doi: 10.1016/j.tjnut.2023.04.010. Epub 2023 Apr 13. PMID 37059395